CLINICAL TRIAL: NCT05269394
Title: A Phase II/III Multicenter Randomized, Double-Blind, Placebo-Controlled Platform Trial of Potential Disease Modifying Therapies Utilizing Biomarker, Cognitive, and Clinical Endpoints in Dominantly Inherited Alzheimer's Disease
Brief Title: Dominantly Inherited Alzheimer Network Trial: An Opportunity to Prevent Dementia. A Study of Potential Disease Modifying Treatments in Individuals With a Type of Early Onset Alzheimer's Disease Caused by a Genetic Mutation (DIAN-TU)
Acronym: DIAN-TU
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH); Accelerating Medicines Partnership (AMP) (Other); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIAN-TU-001 (E2814); The Alzheimer's Association (Other Grant/Funding Number: DIAN TTU-12-243040); U01AG042791 (NIH); 2013-000307-17 (EudraCT Number); R01AG046179 (NIH); REec-2014-0817 (Registry Identifier: Spanish Clinical Studies Registry); The Alzheimer's Association (Other Grant/Funding Number: DIAN-TU Tau-15-347219); GHR Foundation (Other Grant/Funding Number: File 4401); Alzheimer's Association (Other: HDE 18S84914); The Alzheimer's Association (Other Grant/Funding Number: DIAN-TU NG-16-434362); R56AG053267 (NIH); U01AG059798 (NIH); R01AG053267 (NIH); R01AG068319 (NIH); The Alzheimer's Association (Other Grant/Funding Number: DIAN-TU Tau-21822987); The Alzheimer's Association (Other: DIAN-TU OLE-21725093)
Record Dates: First submitted 2022-01-13; First posted 2022-03-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Alzheimers Disease; Dementia; Alzheimers Disease, Familial
Keywords: Alzheimer's; Alzheimer's Disease; Dementia; Mutation; Genetic Mutation; Dominantly Inherited Alzheimer's Disease; Dominantly Inherited Alzheimer Network; Autosomal Dominant Alzheimer's Disease; Early Onset Alzheimer's Disease; DIAN; DIAN-TU; DIAN TU; DIAD
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — lecanemab

STUDY DESIGN:
Intervention Model Description: Interventional
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E2814 plus lecanemab (Experimental): Symptomatic Population (Cohort 1)
  At Week 0, participants will receive open-label lecanemab administered intravenously for the full treatment period.
  At Week 24, participants randomized to E2814 will receive intravenously in a blinded fashion for the remainder of their treatment period.
  Asymptomatic Population (Cohort 2)
  At Week 0, participants randomized to E2814 will receive intravenously in a blinded fashion for the full treatment period.
  At Week 52, all participants will initiate open-label lecanemab administered intravenously for the remainder of their treatment period.
  Interventions: Drug: E2814; Drug: Lecanemab
- Matching placebo (E2814) plus lecanemab (Placebo Comparator): Symptomatic Population (Cohort 1)
  At Week 0, participants will receive open-label lecanemab administered intravenously for the full treatment period.
  At Week 24, participants randomized to E2814 placebo will receive placebo intravenously in a blinded fashion for the remainder of their treatment period.
  Asymptomatic Population (Cohort 2)
  At Week 0, participants randomized to E2814 placebo will receive placebo intravenously in a blinded fashion for the full treatment period.
  At Week 52, all participants will initiate open-label lecanemab administered intravenously for the remainder of their treatment period.
  Interventions: Drug: Lecanemab; Drug: Matching Placebo (E2814)

INTERVENTIONS:
Drug: E2814 — Administered intravenously in a blinded fashion
  Arms: E2814 plus lecanemab
Drug: Lecanemab — Administered intravenously
  Other Names: BAN2401
Drug: Matching Placebo (E2814) — Placebo administered intravenously in a blinded fashion.
  Arms: Matching placebo (E2814) plus lecanemab

SUMMARY:
To assess the safety, tolerability, biomarker, cognitive, and clinical efficacy of investigational products in participants with an Alzheimer's disease-causing mutation by determining if treatment with the study drug improves disease-related biomarkers and slows the rate of progression of cognitive or clinical impairment.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is characterized pathologically by the presence of accumulation of amyloid plaques and tau-containing neurofibrillary tangles (NFTs) in the brain. Amyloid plaques can be detectable within the brain some years before symptoms manifest whereas tau-mediated toxicity has been hypothesized to appear later during the course of disease. Physiologically, tau is predominantly a neuronal microtubule-associated protein that plays a fundamental role in the stabilization of microtubules. Under pathological conditions however, short motifs in the microtubule binding region (MTBR) domains of tau adopt a beta-sheet conformation, inducing self-assembly with other tau molecules that lead to the formation of insoluble aggregates. Insoluble tau is also a feature of a number of different neurodegenerative diseases collectively termed tauopathies. The accumulation of insoluble deposits has been suggested to result in altered distribution and function of organelles to adversely affect neuronal cell function as well as causing synapse loss, ultimately leading to cell death. In AD, evidence also suggests a direct correlation between the number of NFTs found in the brain at postmortem and the degree of dementia observed in subjects with AD at the time of death.

The microtubule-associated protein tau (MAPT) gene is located on chromosome 17 of the human genome. Through alternative splicing, 6 possible tau protein isoforms are expressed from this gene in the adult brain. A number of studies have suggested that pathological forms of tau protein transmit from neuron to neuron in human brain to cause disease, including AD. It has also been reported that tau can form seeds, which when applied extracellularly, can cause the initiation and propagation of intracellular tau aggregation. To form tau seeds, the MTBR of the protein is required. Furthermore, the tau MTBR is important in initiating the tau aggregation process and forming the core of fibrils pathologically associated with disease. Together, these observations suggest that therapeutic intervention with an antibody that binds to the MTBR region of tau in the brain, thereby disrupting tau aggregation may prevent initiation or slow down the neurodegeneration in AD or other tauopathies.

Upcoming Dominantly Inherited Alzheimer Network Trials Unit (DIAN-TU) trials are designed to investigate therapies targeting tau in combination with amyloid as pre-specified in the approved and NIH-funded NexGen Prevention Trial grants. As with other amyloid lowering drug trials, clinical benefit was not definitively demonstrated in the symptomatic population after tau pathology has been established. Determining the role of tau in disease biology and progression is critically important. Based on beneficial effects on amyloid, tau, and neurodegeneration markers associated with amyloid removal in the gantenerumab trial arm in DIAN-TU, the DIAN-TU will now implement amyloid removal treatment in mutation carriers and add placebo- controlled tau treatment arms. The platform trial design is exceptionally well-suited for the investigation of treatments used in combination because of ongoing multiple arms in a single trial and operational platform.

The current DIAN-TU amyloid removal drug arm has been extended to open-label extension (OLE) periods for prior participants. All enrolled participants who opted-in for OLE were unblinded to genetic status and offered open-label gantenerumab treatment. New treatment- naive mutation positive participants will be started on amyloid removal treatment with genetic counseling and testing. Therefore, all participants will be required to be positive for a dominantly inherited Alzheimer's disease (DIAD) mutation and will receive open-label treatment with lecanemab, an investigational amyloid removal drug, in combination with E2814, an anti-tau drug or placebo. Mutation non-carriers will not be enrolled. Specifically, all E2814 blinded drug arm participants will be treated with the lecanemab and randomized to either active E2814 tau therapy, or placebo.

The goal of the study is to investigate potential benefits of anti-tau therapy while anti-amyloid treatment is given as a background therapy. Furthermore, from ethical and participant recruitment perspectives, launching drug trials using amyloid and tau targeting therapies in combination may be essential, as participants and their families have expressed the need to have a drug that changes amyloid disease pathology in addition to being randomized to an investigational anti-tau drug (E2814) with uncertain benefit.

This record represents an analysis study portion of the Master Protocol Research Program (MPRP) under NCT01760005

ELIGIBILITY:
Key Inclusion Criteria:

* Between 18-80 years of age
* Individuals who know they have an Alzheimer's disease-causing mutation.
* Are within -10 to + 10 years of the predicted or actual age of cognitive symptom onset.
* Cognitively normal or with mild cognitive impairment or mild dementia, Clinical Dementia Rating (CDR) of 0-1 (inclusive)
* Fluency in DIAN-TU trial approved language and evidence of adequate premorbid intellectual functioning
* Able to undergo Magnetic Resonance Imaging (MRI), Lumbar Puncture (LP), Positron Emission Tomography (PET), and complete all study related testing and evaluations.
* For women of childbearing potential, if partner is not sterilized, participant must agree to use effective contraceptive measures (hormonal contraception, intra-uterine device, sexual abstinence, barrier method with spermicide).
* Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments.
* Has a Study Partner who in the investigator's judgment is able to provide accurate information as to the subject's cognitive and functional abilities, who agrees to provide information at the study visits which require informant input for scale completion.

Key Exclusion Criteria:

* Significant neurologic disease (other than AD) or psychiatric disease that may currently or during the course of the study affect cognition or participant's ability to complete the study.
* At high risk for suicide, e.g., significant suicidal ideation or attempt within last 12 months. Current stable mild depression or current use of antidepressant medications is not exclusionary.
* History or presence of brain MRI scans indicative of any other significant abnormality
* Substance or alcohol use disorder currently or within the past 1 year
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin or body which would preclude MRI scan.
* History or presence of clinically significant cardiovascular disease, hepatic/renal disorders, infectious disease or immune disorder, or metabolic/endocrine disorders
* Anticoagulants except low dose (≤ 325 mg) aspirin.
* Have been exposed to a monoclonal antibody targeting beta amyloid peptide within the past six months.
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
* Positive urine or serum pregnancy test or plans or desires to become pregnant during the course of the trial.
* Subjects unable to complete all study related testing, including implanted metal that cannot be removed for MRI scanning, required anticoagulation and pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The primary end point is the change from Week 24 to Week 104 and Week 208 in tau PET in the Symptomatic Population (Cohort 1). | Weeks 24, 104, and 208
  To determine whether E2814 is superior to placebo, when each is concurrently administered with lecanemab, in the change from Week 24 to Week 104 (interim analysis) and Week 208 (final analysis) in tau spread as measured by tau PET in the symptomatic population (Cohort 1).

SECONDARY OUTCOMES:
Symptomatic Population (Cohort 1): Key Secondary: Change from Week 24 to Week 208 in Clinical Dementia Scale - Sum of Boxes (CDR-SB). | Weeks 24, 52, 104, 156 and 208
  To determine whether E2814 is superior to placebo, when each is concurrently administered with lecanemab, in change from Week 24 to Week 208 in CDR-SB
  Scores range from 0-18 with lower scores showing better outcomes
Asymptomatic Population (Cohort 2): Key Secondary: Change from Week 0 to Week 104 and Week 208 in CSF ptau217/total tau | Weeks 0, 104 and 208
  To determine whether E2814 is superior to placebo, when each is administered alone and then concurrently with lecanemab, in change from Week 0 to Week 104 (interim analysis) and Week 208 (final analysis) in cerebrospinal fluid (CSF) phosphorylated tau (ptau217)/total tau
Symptomatic Population (Cohort 1): Change from Week 24 to Week 104 and Week 208 in the cognitive composite score | Weeks 24, 52, 76, 104, 128, 156, 180 and 208
Symptomatic Population (Cohort 1): Change from Week 0 to Week 24 in amyloid PET | Week 0 to Week 24
Asymptomatic Population (Cohort 2): Change from Week 0 to Week 52 in CSF ptau217/total tau | Week 0 to Week 52
Symptomatic population (Cohort 1): Change from Week 24 to Week 104 and Week 208 in CSF neurofilament light chain (NfL) | Weeks 24, 104 and 208
Asymptomatic Population (Cohort 2): Change from Week 52 to Week 104 and Week 208 in CSF neurofilament light chain (NfL) | Weeks 52, 104 and 208

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Bateman, MD, Study Director — Washington University School of Medicine
Locations (36):
- United States (12):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - USC Keck School of Medicine, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Kerwin Research Center,, Dallas, Texas
  - University of Washington, Seattle, Washington
- Instituto de Investigaciones Neurologicas Raul Carrea, FLENI, Ciudad Autonoma de Buenos Aire, Argentina
- Australia (2):
  - Neuroscience Research Australia, Randwick, New South Wales
  - Mental Health Research Institute, Melbourne, Victoria
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, Brazil
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill Center for Studies in Aging, Verdun, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec
- Grupo de Neurociencias Sede de la Universidad de Antioquia, Medellín, Colombia
- France (5):
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
- Germany (2):
  - Universitaetsklinikum Tubingen, Tübingen, Baden-Wurttemberg
  - LMU-Campus Grosshadern, Munich, Bavaria
- St Vincent's University Hospital, Dublin, Dublin, Ireland
- Italy (2):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
- University of Tokyo Hospital, Bunkyō City, Tokyo-To, Japan
- Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez, Mexico City, Mexico City, Mexico
- Brain Research Center, Amsterdam, Netherlands
- University of Puerto Rico, School of Medicine, San Juan, Puerto Rico, Puerto Rico
- Hospital Clínic I Provincial de Barcelona, Barcelona, Barcelona, Spain
- The National Hospital for Neurology and Neurosurgery, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to DIAN-TU trial data will follow the DIAN-TU data access policy, which complies with the guidelines established by the Collaboration for Alzheimer's Prevention [CAP REF].

REFERENCES:
- [Background] Jack CR Jr, Knopman DS, Jagust WJ, Petersen RC, Weiner MW, Aisen PS, Shaw LM, Vemuri P, Wiste HJ, Weigand SD, Lesnick TG, Pankratz VS, Donohue MC, Trojanowski JQ. Tracking pathophysiological processes in Alzheimer's disease: an updated hypothetical model of dynamic biomarkers. Lancet Neurol. 2013 Feb;12(2):207-16. doi: 10.1016/S1474-4422(12)70291-0. PMID 23332364
- [Background] Fitzpatrick AWP, Falcon B, He S, Murzin AG, Murshudov G, Garringer HJ, Crowther RA, Ghetti B, Goedert M, Scheres SHW. Cryo-EM structures of tau filaments from Alzheimer's disease. Nature. 2017 Jul 13;547(7662):185-190. doi: 10.1038/nature23002. Epub 2017 Jul 5. PMID 28678775
- [Background] Falcon B, Zhang W, Murzin AG, Murshudov G, Garringer HJ, Vidal R, Crowther RA, Ghetti B, Scheres SHW, Goedert M. Structures of filaments from Pick's disease reveal a novel tau protein fold. Nature. 2018 Sep;561(7721):137-140. doi: 10.1038/s41586-018-0454-y. Epub 2018 Aug 29. PMID 30158706
- [Background] Kopeikina KJ, Hyman BT, Spires-Jones TL. Soluble forms of tau are toxic in Alzheimer's disease. Transl Neurosci. 2012 Sep;3(3):223-233. doi: 10.2478/s13380-012-0032-y. PMID 23029602
- [Background] Braak H, Braak E. Neuropathological stageing of Alzheimer-related changes. Acta Neuropathol. 1991;82(4):239-59. doi: 10.1007/BF00308809. PMID 1759558
- [Background] Goedert M, Spillantini MG. Propagation of Tau aggregates. Mol Brain. 2017 May 30;10(1):18. doi: 10.1186/s13041-017-0298-7. PMID 28558799
- [Background] Falcon B, Cavallini A, Angers R, Glover S, Murray TK, Barnham L, Jackson S, O'Neill MJ, Isaacs AM, Hutton ML, Szekeres PG, Goedert M, Bose S. Conformation determines the seeding potencies of native and recombinant Tau aggregates. J Biol Chem. 2015 Jan 9;290(2):1049-65. doi: 10.1074/jbc.M114.589309. Epub 2014 Nov 18. PMID 25406315
- [Background] Barghorn S, Zheng-Fischhofer Q, Ackmann M, Biernat J, von Bergen M, Mandelkow EM, Mandelkow E. Structure, microtubule interactions, and paired helical filament aggregation by tau mutants of frontotemporal dementias. Biochemistry. 2000 Sep 26;39(38):11714-21. doi: 10.1021/bi000850r. PMID 10995239
- [Background] von Bergen M, Friedhoff P, Biernat J, Heberle J, Mandelkow EM, Mandelkow E. Assembly of tau protein into Alzheimer paired helical filaments depends on a local sequence motif ((306)VQIVYK(311)) forming beta structure. Proc Natl Acad Sci U S A. 2000 May 9;97(10):5129-34. doi: 10.1073/pnas.97.10.5129. PMID 10805776
- [Background] von Bergen M, Barghorn S, Li L, Marx A, Biernat J, Mandelkow EM, Mandelkow E. Mutations of tau protein in frontotemporal dementia promote aggregation of paired helical filaments by enhancing local beta-structure. J Biol Chem. 2001 Dec 21;276(51):48165-74. doi: 10.1074/jbc.M105196200. Epub 2001 Oct 17. PMID 11606569
- [Background] Salloway S, Farlow M, McDade E, Clifford DB, Wang G, Llibre-Guerra JJ, Hitchcock JM, Mills SL, Santacruz AM, Aschenbrenner AJ, Hassenstab J, Benzinger TLS, Gordon BA, Fagan AM, Coalier KA, Cruchaga C, Goate AA, Perrin RJ, Xiong C, Li Y, Morris JC, Snider BJ, Mummery C, Surti GM, Hannequin D, Wallon D, Berman SB, Lah JJ, Jimenez-Velazquez IZ, Roberson ED, van Dyck CH, Honig LS, Sanchez-Valle R, Brooks WS, Gauthier S, Galasko DR, Masters CL, Brosch JR, Hsiung GR, Jayadev S, Formaglio M, Masellis M, Clarnette R, Pariente J, Dubois B, Pasquier F, Jack CR Jr, Koeppe R, Snyder PJ, Aisen PS, Thomas RG, Berry SM, Wendelberger BA, Andersen SW, Holdridge KC, Mintun MA, Yaari R, Sims JR, Baudler M, Delmar P, Doody RS, Fontoura P, Giacobino C, Kerchner GA, Bateman RJ; Dominantly Inherited Alzheimer Network-Trials Unit. A trial of gantenerumab or solanezumab in dominantly inherited Alzheimer's disease. Nat Med. 2021 Jul;27(7):1187-1196. doi: 10.1038/s41591-021-01369-8. Epub 2021 Jun 21. PMID 34155411
- [Background] Sandusky-Beltran LA, Sigurdsson EM. Tau immunotherapies: Lessons learned, current status and future considerations. Neuropharmacology. 2020 Sep 15;175:108104. doi: 10.1016/j.neuropharm.2020.108104. Epub 2020 Apr 28. PMID 32360477
- See also: Expanded registry — http://www.dianexr.org/